CLINICAL TRIAL: NCT05435131
Title: Evaluation of Interleukin (IL)-38, IL-36-gamma, IL-17 and Matrix Metalloproteinase-9 Levels in Gingival Crevicular Fluid, Saliva and Serum for Periodontal Health, Gingivitis and Periodontitis
Brief Title: Evaluation of Biomarkers Levels in Gingival Crevicular Fluid, Saliva and Serum for Different Periodontal Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hilal Korkmaz, Research Assistant, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Hkorkmaz
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Mouth Diseases; Periodontal Inflammation; Periodontal Diseases
MeSH Terms: conditions — Mouth Diseases; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: According to full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL),bleeding on probing (BOP), gingival index (GI) and plaque index (PI) samples of GCF, saliva and serum were obtained from 90 systemically healthy non-smoker individuals with stage II grade B (P1, n=9), stage III grade B (P2, n=11) , stage III grade C (n=10), gingivitis (G, n=30) and healthy periodontium (S, n=30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Periodontal Health (Experimental): Full-mouth clinical periodontal measurements recorded and GCF, saliva serum obtained.
  Interventions: Diagnostic Test: GCF obtaining; Diagnostic Test: Saliva Obtaining; Diagnostic Test: Serum obtaining
- Gingivitis (Experimental): Full-mouth clinical periodontal measurements recorded and GCF, saliva serum obtained.
  Interventions: Diagnostic Test: GCF obtaining; Diagnostic Test: Saliva Obtaining; Diagnostic Test: Serum obtaining
- Stage II grade B Periodontitis (Experimental): Full-mouth clinical periodontal measurements recorded and GCF, saliva serum obtained.
  Interventions: Diagnostic Test: GCF obtaining; Diagnostic Test: Saliva Obtaining; Diagnostic Test: Serum obtaining
- Stage III grade B Periodontitis (Experimental): Full-mouth clinical periodontal measurements recorded and GCF, saliva serum obtained.
  Interventions: Diagnostic Test: GCF obtaining; Diagnostic Test: Saliva Obtaining; Diagnostic Test: Serum obtaining
- Stage III grade C Periodontitis (Experimental): Full-mouth clinical periodontal measurements recorded and GCF, saliva serum obtained.
  Interventions: Diagnostic Test: GCF obtaining; Diagnostic Test: Saliva Obtaining; Diagnostic Test: Serum obtaining

INTERVENTIONS:
Diagnostic Test: GCF obtaining — GCF obtaining: 2 GCF samples, 1 from the interproximal surface of 2 different teeth that bleeding on probing(-), were taken from each participant
Diagnostic Test: Saliva Obtaining — Saliva obtaining: 1,5 ml unstimulated whole saliva collected from each participant
Diagnostic Test: Serum obtaining — Serum obtaining : 8 ml of venous blood was collected from each participant and collecting blood centrifuged to obtain serum

SUMMARY:
The aim of this study is; detection of interleukin(IL)-38, IL-36 gamma(γ) , IL-17 and matrix metalloproteinase(MMP)-9 levels in gingival crevicular fluid (GCF), saliva and serum samples of periodontally healthy, gingivitis and periodontitis patients and the possible correlation between these values and clinical parameters of periodontal diseases. Materials and methods: Samples were obtained from 90 systemically healthy non-smoker individuals with periodontitis (P, n=30), gingivitis(G, n=30) and healthy periodontium (S, n=30). Full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were also recorded. Enzyme-linked immunosorbent assay (ELISA) was used to determine IL-38, IL-36γ, IL-17 and MMP-9 levels in the biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (The determination of healthy volunteers will be based on the statements of the patients in the anamnesis. No additional examinations will be made.)
* At least twenty permanent teeth in the mouth
* Non-smoker
* No medication for continuous use
* Those who have not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 6 months.
* Not in pregnancy or lactation period.
* For the periodontitis group that has not received periodontal treatment in the last 6 months

Exclusion Criteria:

* Any oral or systemic disease
* Regularly using a systemic medication
* During pregnancy or lactation
* Received periodontal treatment within the last 6 months.
* Those who received antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months
* Smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Levels of Interleukin-38 (pg/ml) in GCF, saliva and serum fluid | 24 hours after taking the clinical measurements at the first visit
Levels of Interleukin-36 gamma (pg/ml) in GCF, saliva and serum fluid | 24 hours after taking the clinical measurements at the first visit

SECONDARY OUTCOMES:
Levels of Interleukin-17 (pg/ml) in GCF, saliva and serum fluid | 24 hours after taking the clinical measurements at the first visit
Levels of Matrix Metalloproteinase-9 (ng/ml) in GCF, saliva and serum fluid | 24 hours after taking the clinical measurements at the first visit

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Faculty of Dentistry, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF